CLINICAL TRIAL: NCT03823053
Title: The Effect of Core Stabilization Training on Respiratory Parameters, Peripheral Muscle Strength, Balance, Functional Capacity and Quality of Life in Children With Adolescent Idiopathic Scoliosis
Brief Title: The Effect of the Core Stabilization Training on Respiratory Parameters , Functional Capacity and Balance in Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BVUsyildirim01
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent idiopathic scoliosis; Scoliosis; Core Stabilization Training; Exercise Training; Pulmonary Function Test; 6 - Minute Walk Test; Peripheral Muscle Strength; Balance with Biodex; Quality of Life
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group will be given home based traditional scoliosis exercise training for 8 weeks, 5 days a week for 30 minutes. The content of the physiotherapy program; posture, interscapular muscle strengthening, stretching and lateral flexion exercises are formed.
  Interventions: Other: Home Based Traditional Scoliosis Exercise
- Training Group (Experimental): In addition to home based traditional scoliosis exercise, the training group will also receive core stabilization exercise training for 8 weeks, 5 days a week, for 30 minutes. Core stabilization training; exercises for 2 muscle systems that contribute to spinal stability are given. The first one is the "local system" muscles; multifidus, transversus abdominis, diaphragm and pelvic floor muscles. The second, the "global system" includes large superficial muscles, such as erector spines, rectus abdominis, internal and external obliques, quadratus lumborum, gluteus maximus, and latissimus dorsi.
  Interventions: Other: Home Based Traditional Scoliosis Exercise; Other: Home Based Core Stabilization Training

INTERVENTIONS:
Other: Home Based Traditional Scoliosis Exercise — Program will include posture exercises, strengthening exercises of interscapular muscle and limb, diaphragmatic breathing exercises and stretching exercises for lumbar extensor, hip flexor, hamstring, pectoral muscles. Exercises will be applied 1 sets of 10 repetitions and once a day.
Other: Home Based Core Stabilization Training — Program will include posture exercises, strengthening exercises of interscapular muscle and limb, diaphragmatic breathing exercises and stretching exercises for lumbar extensor, hip flexor, hamstring, pectoral muscles. In addition, the training group received core stabilization exercises for multifidus, transversus abdominis, diaphragm,erector spines, rectus abdominis, internal and external obliques, quadratus lumborum, gluteus maximus, and pelvic floor muscles.Exercises will be applied 1 sets of 10 repetitions and once a day.
  Arms: Training Group

SUMMARY:
The vertebral column is a structure that transfers the weight of the head and torso to the lower extremity, provides trunk movements and protects the spinal cord.A three dimensional deformity involving lateral flexion of the vertebrae in the frontal plane at 10 ° and above, including axial rotation and physiologic flexion (hypokyphosis) components in the sagittal plane, is defined as scoliosis. Adolescent idiopathic scoliosis (AIS) is a type of idiopathic scoliosis that occurs in the period from the onset of puberty (up to 10 years) until the closure of growth plates.

Scoliosis is caused by postural, balance and neuromotor disorders as a primary cause of impaired sensory integrity, proprioceptive feedback deficits, secondary lung problems, organ disorders and pain. In addition, the quality of life in these individuals is also seen to decrease.Children with adolescent idiopathic scoliosis have inadequate respiratory function and a decrease in functional capacity. At the same time, these children show muscle weakness in certain parts of the body.

The aim of this study was to investigate the relationship between home based core stabilization training, respiratory parameters, peripheral muscle strength, balance, functional capacity and quality of life in individuals with young scoliosis. The investigators suggest that the addition of core stabilization training to children with mild and moderate adolescent idiopathic scoliosis will produce good results.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent Idiopathic Scoliosis diagnosis

Exclusion Criteria:

* Documented diagnosis any of cardiopulmonary, neurological, orthopedic or mental disorders which may affect the assessments results.
* Subjects previously undertaken any of spinal surgeries.
* Subjects involved in exercise training 3 or more days a week.

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline Forced Vital Capacity (FVC) at 8 weeks | Eight weeks
Change from baseline Forced Expiratory volume in 1 second (FEV1)at 8 weeks | Eight weeks
Change from baseline Peripheral Muscle strength at 8 weeks | Eight weeks
Change from baseline Balance at 8 weeks | Eight weeks
Change from baseline distance covered in Six- Minute Walk Test at 8 weeks | Eight weeks

SECONDARY OUTCOMES:
Change from baseline axial trunk rotation (ATR) | Eight weeks
  Measurements will be applied with Bunnell Scoliometer by physiotherapist.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Eyüp, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yildirim S, Ozyilmaz S, Elmadag NM, Yabaci A. Effects of Core Stabilization Exercises on Pulmonary Function, Respiratory Muscle Strength, Peripheral Muscle Strength, Functional Capacity, and Perceived Appearance in Children With Adolescent Idiopathic Scoliosis: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2022 Aug 1;101(8):719-725. doi: 10.1097/PHM.0000000000001984. Epub 2022 Feb 2. PMID 35859288